CLINICAL TRIAL: NCT00409903
Title: The Effect of Eprosartan on Vasoactive Hormones and Renal Tubular Function in Healthy Humans.
Brief Title: The Effect of Eprosartan on Hormones and Kidney Function in Healthy Humans.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: MED.RES.HOS.2006.02.HV
Record Dates: First submitted 2006-12-10; First posted 2006-12-12 (Estimated); Last update posted 2007-09-14 (Estimated); Status verified 2007-09

CONDITIONS: Healthy
MeSH Terms: interventions — eprosartan

INTERVENTIONS:
Drug: Eprosartan

SUMMARY:
We, the investigators at Holstebro Hospital, want to test the hypothesis that eprosartan reduces the activity of the sympathetic nervous system in healthy individuals - during baseline conditions and after activation of the sympathetic nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* Age 18 - 65 years.
* Body mass index less or equal to 30 kg/m2.
* Women must use oral hormonal anticonception, use intrauterine anticonceptive device, be sterilized/hysterectomized or be postmenopausal.

Exclusion Criteria:

* History or clinical signs of heart, lung, kidney, or endocrine organ disease.
* Abnormal biochemical screening of the blood regarding: B-hemoglobin, P-sodium, P-potassium, P-creatinine, P-albumin, P-bilirubin, P-alanine aminotransferase, P-alkaline phosphatase, P-cholesterol, and B-glucose.
* Abnormal screening of the urine regarding: albumin and glucose
* Malignant disease.
* Known arterial hypertension or measured 24 hour blood pressure above 135 mmHg systolic or 85 mmHg diastolic.
* Alcohol abuse.
* Smoking.
* Drug use or abuse.
* Known intolerance or allergy to eprosartan or sodium nitroprusside.
* Blood donation within 1 month of the start of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2006-11

PRIMARY OUTCOMES:
Heart rate
Fractional sodium excretion
Plasma levels of noradrenaline

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, MD, professor, Study Chair — Department of Medical Research, Holstebro Hospital, Denmark
Locations (1):
- Department of Medical Research, Holstebro Hospital, Holstebro, Denmark